CLINICAL TRIAL: NCT02827110
Title: Tracheal Intubation in Patient With Semi-rigid Collar Immobilization of the Cervical Spine: A Comparison of Fiberoptic Bronchoscope Assisted With Pentax-airway Scope and Fiberoptic Bronchoscope Alone
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ajou University School of Medicine (Other)
Responsible Party: Principal Investigator, yun jeong chae, Associate Professor, Ajou University School of Medicine
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: AJIRB-MED-DE2-16-060
Record Dates: First submitted 2016-06-16; First posted 2016-07-11 (Estimated); Last update posted 2017-06-28 (Actual); Status verified 2017-06

CONDITIONS: Cholecystitis
MeSH Terms: conditions — Cholecystitis

ARMS (2):
- fiberoptic bronchoscope (Active Comparator): Tracheal intubation in patients with semi-rigid collar immobilization of the cervical spine using fiberoptic bronchoscope
  Interventions: Device: fiberoptic bronchoscope; Procedure: semi-rigid collar
- fiberoptic bronchoscope with pentax-AWS (Experimental): Tracheal intubation in patients with semi-rigid collar immobilization of the cervical spine using fiberoptic bronchoscope with pentax-AWS
  Interventions: Device: fiberoptic bronchoscope; Device: pentax-airway scope; Procedure: semi-rigid collar

INTERVENTIONS:
Device: fiberoptic bronchoscope — Tracheal intubation using fiberoptic bronchoscope
Device: pentax-airway scope — Tracheal intubation using pentax-AWS
  Arms: fiberoptic bronchoscope with pentax-AWS
Procedure: semi-rigid collar — semi-rigid collar immobilization of the cervical spine

SUMMARY:
A semi-rigid cervical collar is recommended for immobilization of the cervical spine in patients with cervical spine injury. It has been suggested that a reduction in mouth opening is the major contributing factor to the deterioration in the glottic view obtained. Fiberoptic intubation is among the most versatile techniques for managing both the anticipated and the unanticipated difficult airway. Recently, combination of fiberoptic bronchoscope with videolaryngoscope has been suggested to permit visual control of the passage of the tube over the fibrescope into the laryngeal inlet. The aim of this study is to compare the intubation time and ease of intubation between fiberoptic bronchoscope alone and bronchoscope with pentax airwayscope.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiologist physical status class I, II

Exclusion Criteria:

* uncontrolled or limited cardiovascular disease
* abnormality of airway
* necessity for rapid sequence induction
* BMI > 30

Ages: 20 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Actual)
Dates: Start 2016-06 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
time to intubation | Time from device passing the mouth until confirmation of tracheal intubation by bronchoscope will be measured, about 2 minutes

SECONDARY OUTCOMES:
ease of intubation | Numeric rating scale will be assessed by practioner of fiberoptic bronchoscope for intubation immediately after intubation.
  Numeric rating scale 0-10 (0:easy without any difficulty, 10: impossible to intubate)

CONTACTS AND LOCATIONS:
Locations (1):
- Ajou University School of Medicine, Suwon, Gyeonggi-do, South Korea

REFERENCES:
- [Derived] Kim DH, Yoo JY, Ha SY, Chae YJ. Comparison of the paediatric blade of the Pentax-AWS and Ovassapian airway in fibreoptic tracheal intubation in patients with limited mouth opening and cervical spine immobilization by a semi-rigid neck collar: a randomized controlled trial. Br J Anaesth. 2017 Nov 1;119(5):993-999. doi: 10.1093/bja/aex272. PMID 28981579